CLINICAL TRIAL: NCT04570592
Title: Granisetron vs Granisetron and Dexamethasone on the Reduction of Postoperative Nausea and Vomiting After Caesarean Section With Intrathecal Morphine: A Randomized Controlled Trial
Brief Title: Granisetron vs Granisetron and Dexamethasone on the Reduction of Postoperative Nausea and Vomiting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Farah Nasuha Mohd Daut, Trainee Anaesthetist, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/JEPeM/1809426
Record Dates: First submitted 2020-09-19; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: PONV
Keywords: Caesarean; Morphine; Granisetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Granisetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granisetron (Placebo Comparator): Granisetron 1 mg (1ml) + Normal saline 1ml
  Interventions: Drug: Granisetron 1 Mg/mL Intravenous Solution
- Granisetron and Dexamethasone (Experimental): Granisetron 1mg (1ml) + Dexamethasone 4mg (1ml)
  Interventions: Drug: Granisetron 1 Mg/mL Intravenous Solution And Dexamethasone 4mg

INTERVENTIONS:
Drug: Granisetron 1 Mg/mL Intravenous Solution And Dexamethasone 4mg — Comparing PONV incidences in both arms
  Other Names: Treatment group
  Arms: Granisetron and Dexamethasone
Drug: Granisetron 1 Mg/mL Intravenous Solution — Comparing PONV incidences in both arms
  Arms: Granisetron

SUMMARY:
Intrathecal morphine (ITM) has proven to be excellent in reducing postoperative pain. However, its use has commonly been associated with the occurrence of postoperative nausea and vomiting (PONV). In recent years, the combination therapy of antiemetics comprising of a serotonin receptor antagonist and corticosteroid has been implemented to diminish the occurrence of PONV. Despite being routinely used, the evidence in the efficacy of this combination in parturients are conflicting and lacking. In this study, we wish to compare the efficacy between the combination therapy of granisetron plus dexamethasone versus granisetron alone on the occurrence of postoperative nausea and vomiting (PONV) in 126 parturients undergoing elective Caesarean delivery supplemented with intrathecal morphine.

DETAILED DESCRIPTION:
126 parturients aged between 18 and 45 years old who falls within the American Society of Anaesthesiology (ASA) physical status I and II undergoing Caesarean deliveries from the 1st of October 2020 till the 1st of April 2021 will be enrolled. Informed and written consent shall be obtained on recruitment.

Subjects will be randomised using a computer-generated randomisation software using block size 3 into 2 groups; group A and group B each consisting of 63 subjects. The order of interventions within each block was random as determined by computer random number generator. This technique was chosen to ensure similar numbers of patients in each group at any point during the study. Both patients and the assessors of PONV which is the Acute Pain Service (APS) team will be blinded.

Patients are subjected to fasting 6 hours prior to surgery with clear fluid allowed up to 2 hours before surgery. Intravenous (IV) metaclopromide 10mg, IV ranitidine 50mg and mist sodium citrate 30 mls will be administered as part of the acid aspiration prophylaxis. Standard monitoring with continuous noninvasive blood pressure monitoring (NIBP), electrocardiogram (ECG), respiratory rate and pulse oximetry (SpO2) will be implemented throughout anaesthesia.

Ringer's lactate solution 10ml/kg will be infused for coloading to mitigate hypotension post spinal anaesthesia. Spinal anaesthesia will be administered in the upright position, implementing a height-based dose for heavy bupivacaine 0.5% administration. Based on the subject's height, those who are less than 150cm, 151-154cm and those who are more than 155cm will receive 1.5mls, 1.7mls and 1.9mls heavy bupivacaine 0.5% (AstraZeneca) respectively. Fentanyl 15-20 mcg and morphine 0.1 mg are added to supplement the spinal anaesthesia.

On the completion of spinal anaesthesia, 4 mg of dexamethasone will be administered to parturients in group A while group B received 1ml of normal saline injected intravenously. 1mg of IV granisetron will be administered to both groups of subjects after cord clamping. These drugs will be given by the anaesthetist administering the spinal anaethesia. The anaesthetist in charge is not blinded as this is of paramount importance in ensuring patients safety should any complication arises during the delivery of anaesthesia.

Post surgery, subjects will be monitored in the recovery area for an hour. To supplement ITM as the postoperative analgesia, tablet paracetamol 1g qid and voltaren 50mg tds will be provided to patients postoperatively. The use of opioid is avoided during the first 24 hours of intrathecal morphine administration. Patients will be monitored for complications of ITM for 24 hours and assessments will be carried out by the APS team which include an anaesthetic medical officer and 2 staff nurses.

Assessments are made at 1 hour post surgery, 4 hourly for 12 hours post surgery up to 24 hours after surgery. Episodes of nausea, retching and vomiting will be elicited by direct questioning and recorded at each assessors' visit. Nausea is described as an unpleasant sensation related to the urge to vomit. Retching is defined as an involuntary effort to vomit but without the expulsion of the gastric contents, while vomiting is the when expulsion of gastric contents occur.

The requirement of rescue antiemetics at each time interval will also be documented. Rescue antiemetic is given when a patient developed one or more episodes of vomiting. IV ondansetron 4 mg is given to group A while either IV dexamethasone 4mg or iv ondansetron is given to group B. Subsequent requirement of antiemetics will be decided based on the anaesthetist discretion.

Sample size is calculated based the assumption that the combination of a serotonin receptor antagonist with a corticosteroid would be superior than its monotherapy and thus, the addition of dexamethasone to granisetron would reduce the incidence of PONV from 20% to 3.3%. From the calculation using PS software, the sample required for each group is 57, and with the additional 10% for dropout rate, this study required 63 patients in each group, giving a total of 126 patients.

Data analysis will be performed using SPSS version 27 for MAC. The incidences of nausea, retching, vomiting and the use of rescue antiemetic will be analysed using Chi-Square test. Data is presented as percentage and a p-value of <0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) I-II category
* 2 risks factors or more for PONV according to Apfel Score.

Exclusion Criteria:

* Unfit for spinal anaesthesia.
* Coagulopathy
* Uncorrected hypovolemia
* Indeterminate neurologic disease
* Infection at site of injection
* Raised intracranial pressure(ICP)
* Morbidly obese patients, BMI> 40 kg/m2 according to ICD-10 (International Statistical Classification of Diseases 10)
* Patients allergic towards morphine.
* Contraindicated for antiemetics use
* Granisetron: allergy towards Granisetron, prolonged QT interval
* Ondansetron: allergy towards ondansetron, prolonged QT interval
* Dexamethasone: allergy towards Dexamethasone, uncontrolled Diabetes Mellitus (DM).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients
Enrollment: 126 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the incidence of post operative nausea and vomiting (PONV) | From 1 to 24 hour post operatively
  To compare the incidence of nausea, retching and vomiting at 1 hour, 4 hourly for 12 hours and at 24 hours postoperatively between parturients receiving combination therapy of Granisetron plus Dexamethasone versus that of Granisetron alone

SECONDARY OUTCOMES:
Comparing the requirement of rescue antiemetic between both groups | From 1 to 24 hour post operatively
  To compare the requirement of rescue antiemetic between 1 hour, 4 hourly for 12 hours and at 24 hours postoperatively between parturients receiving combination therapy of Granisetron plus Dexamethasone versus that of Granisetron alone

CONTACTS AND LOCATIONS:
Overall Officials: Farah Nasuha Mohd Daut, Principal Investigator — Universiti Sains Malaysia, Health Campus, Kubang Kerian, Kelantan
Locations (1):
- Universiti Sains Malaysia, Health Campus, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD will be considered for sharing if the data is to be used for related studies.

REFERENCES:
- [Background] Gwirtz KH, Young JV, Byers RS, Alley C, Levin K, Walker SG, Stoelting RK. The safety and efficacy of intrathecal opioid analgesia for acute postoperative pain: seven years' experience with 5969 surgical patients at Indiana University Hospital. Anesth Analg. 1999 Mar;88(3):599-604. doi: 10.1097/00000539-199903000-00026. PMID 10072014
- [Background] Sfeir S, Mansour N. Post operative analgesia with intrathecal morphine. Middle East J Anaesthesiol. 2005 Feb;18(1):133-9. PMID 15830768
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Result] Abouleish E, Rawal N, Fallon K, Hernandez D. Combined intrathecal morphine and bupivacaine for cesarean section. Anesth Analg. 1988 Apr;67(4):370-4. PMID 3354872